CLINICAL TRIAL: NCT01184157
Title: Randomized Trial of Home Versus Clinic-based Screening for Sexually Transmitted Infections in Long-Acting Reversible Contraceptive Users
Brief Title: Randomized Trial of Home Versus Clinic-based Screening for Sexually Transmitted Infections
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Washington University School of Medicine (Other)
Responsible Party: Jeffrey Peipert, MD PhD, Washington University School of Medicine
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Screening
Other Study IDs: 07-0256
Record Dates: First submitted 2010-08-17; First posted 2010-08-18 (Estimated); Last update posted 2010-08-18 (Estimated); Status verified 2010-08

CONDITIONS: Chlamydia; Gonorrhea
MeSH Terms: conditions — Chlamydia Infections; Gonorrhea

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Home (Experimental): Home-based STI screening using self-obtained vaginal swabs and postal return of samples.
  Interventions: Behavioral: Home screening
- Clinic (Active Comparator): Receive STI screening in a clinical setting such as a private physician or clinic.
  Interventions: Behavioral: Clinic screening

INTERVENTIONS:
Behavioral: Home screening
  Arms: Home
Behavioral: Clinic screening
  Arms: Clinic

SUMMARY:
This study randomizes women using long-acting reversible methods of contraception to home-based STD screening through the mail compared to screening available in a clinical setting. We hypothesize that women randomized to home-based screening will be more likely to complete screening.

ELIGIBILITY:
Inclusion Criteria:

* Participant in Contraceptive CHOICE cohort study
* Using a long-acting reversible method of contraception
* Completed baseline clinical survey in the Contraceptive CHOICE cohort study

Exclusion Criteria:

* Living outside the United States at time of annual STI screening

Ages: 14 Years to 45 Years | Sex: Female
Age Groups: Child, Adult

PRIMARY OUTCOMES:
Number of tests received

CONTACTS AND LOCATIONS:
Overall Officials: Jeffrey Peipert, MD, PhD, Principal Investigator — Washington University School of Medicine
Locations (1):
- Washington University School of Medicine, St Louis, Missouri, United States

REFERENCES:
- [Derived] Graseck AS, Secura GM, Allsworth JE, Madden T, Peipert JF. Home compared with clinic-based screening for sexually transmitted infections: a randomized controlled trial. Obstet Gynecol. 2010 Dec;116(6):1311-1318. doi: 10.1097/AOG.0b013e3181fae60d. PMID 21099596